CLINICAL TRIAL: NCT05827419
Title: Hearing and Balance Disorders in Peripheral Neuropathy
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit participants
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: TM001
Record Dates: First submitted 2018-06-25; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2018-10

CONDITIONS: Charcot-Marie-Tooth Disease
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and buccal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The long term goal of this proposal is to precisely characterize the auditory and vestibular abilities of children with Charcot-Marie-Tooth (CMT) and how these abilities evolve during the progression of the disorder. This information will be used to refine the management methods for hearing loss and vestibular disorders in these patients. Given that the phenotypic severity is variable within the CMT patient population, we predict that not all CMT patients will present with auditory and vestibular dysfunction. We will therefore collect specimens (i.e., buccal swabs and saliva) from study participants so that their DNA can be isolated and used to determine the genetic basis for auditory and vestibular dysfunction in peripheral neuropathies.

DETAILED DESCRIPTION:
Aim #1: Evaluate the prevalence of auditory and vestibular disorders in children diagnosed with Charcot-Marie-Tooth.

We hypothesize that a significant number of children with Charcot-Marie-Tooth (CMT) will develop auditory and vestibular neuropathies, due to the progression of the disorder. We will examine the characteristics of auditory and vestibular abilities of children and how these relate to the type of CMT.

Aim #2: Examine the progression of hearing and vestibular abilities during the course of the disorder.

We hypothesize that the hearing and vestibular abilities of some children with CMT will deteriorate with time. We will repeat the auditory and vestibular testing on a yearly basis to precisely describe the progression of these abilities.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Charcot-Marie Tooth

Exclusion Criteria:

-

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults between the ages of 5 and 21 years diagnosed with Charcot-Marie-Tooth will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of auditory disorders in children diagnosed with Charcot-Marie-Tooth Characteristics. | 2 years
  We will evaluate how many children with CMT have present hearing loss. The presence of hearing loss will be based on the results of the following tests (passed or failed): otoacoustic emissions, auditory brainstem responses, auditory event related potentials, audiometry and speech perception
Prevalence of vestibular disorders in children diagnosed with Charcot-Marie-Tooth | 2 years
  We will evaluate how many children with CMT have present vestibular disorder. The presence of vestibular disorder will be based on the results of the following test (passed or failed): video head impulse test
Progression of hearing loss | 2 years
  We will follow subjects longitudinally to evaluate the progression of hearing loss. The degree of hearing loss will be monitor over time to evaluate if changes are noticed.
  All tests listed in Outcome 1 will be repeated and compared to initial values to define the presence or absence of changes in the degree of hearing loss.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Morlet, PhD, Principal Investigator — Nemours
Locations (1):
- Nemours, Wilmington, Delaware, United States